CLINICAL TRIAL: NCT03323268
Title: Validation of End-tidal CO2 for Transplumonary Blood Flow Monitoring During PVA-ECMO
Brief Title: Use of Exhaled Carbon Dioxyde for Monitoring the Native Cardiac Function During Mechanical Circulatory Support With Venoarterial By-pass in Intensive Care Unit
Acronym: CAPNOECMO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9653
Record Dates: First submitted 2016-07-12; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2016-07

CONDITIONS: Residual Cardiac Output During PVA-ECMO
Keywords: Intensive care; Cardiogenic shock; Peripheral veno-arterial extracorporeal membrane oxygenation; Left ventricular overload; Native cardiac output; Pulmonary artery blood flow; End-tidal carbon dioxide; Swan Ganz catheter; Blood gaz
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: PetCO2 monitoring — CO2 analyzer on ventilator expiratory lane. On-line, continuous, and noninvasive monitor. Routine use in anesthesia and intensive care units.

SUMMARY:
Cardiogenic shock, the most severe form of acute heart failure, is a critical situation where the body cells lack of oxygen because of cardiac dysfunction. The failure of pharmacological therapy to maintain adequate perfusion has led to attempts to improve the circulation by the use of mechanical circulatory support devices. Peripheral veno-arterial support (PVA-ECMO) is the most frequently used device. It consists of extracorporeal circulatory support. Venous blood is aspirated via the right atrium and reinjected into the descending aorta via the femoral artery. As a consequence of this by-pass, pulmonary artery flow and residual left ventricle ejection can fall drastically until zero in the most severe patients. A minimal transpulmonary blood flow is crucial to avoid left heart cavities and pulmonary artery and left heart cavities thrombosis. The gold standard technique to monitor transpulmonary blood flow is right-heart cavities catheterism (Swan-Ganz catheter) but it represents major limits: invasive technique, limited duration of utilization because of septic risk, physical limit of flow measurement (under 1 liter/minute). End-tidal pressure carbon dioxide (Pet CO2) monitoring (or capnography) is a routine and non-invasive measure in ventilated patients. Previous studies have shown that changes in PetCO2 can measure changes in cardiac output in anesthetized patients and that PetCO2 is a useful index of pulmonary artery blood flow during separation from cardiopulmonary bypass. The aim of this study is to demonstrate that PetCO2 is correlated to transpulmonary blood flow in patients under PVA-ECMO and that exhaled CO2 can provide an on-line, continuous, and noninvasive monitor of residual outflow from the heart during PVA-ECMO.

DETAILED DESCRIPTION:
Settings

This prospective study is conducted since January 2016 in our tertiary ICU and has been approved by our hospital's institutional review board. Informed consent will be obtained from all patients or their surrogates.

Hemodynamic is monitored via a radial arterial catheter for continuous blood pressure monitoring, a pulmonary artery catheter (Swan-Ganz CCOmbo® CCO/SvO2, Edwards Lifesciences) inserted through the superior vena cava (jugular intern or subclavian vein) and transoesophageal echocardiography (TOE) at PVA-ECMO implantation or at operator discretion.

ECMO circuit settings and patients management under ECMO

PVA-ECMO consist of polyvinyl chloride tubing with a membrane oxygenator (PH.I.S.I.O and EOS; Sorin Group, Clamart, France), a centrifugal pump (Stockert; Sorin Group), and percutaneous or surgically inserted arterial and venous femoral cannulae (Fem-Flex and Fem-Track, Edwards Life- sciences, Guyancourt, France) with or without an additional 7 F cannula inserted distally into the femoral artery to prevent lower limb ischemia. An oxygen-air blender (Sechrist Industries, Anaheim, CA) ventilate the membrane oxygenator. Unfractionated heparin is administrated to maintain an activated partial thromboplastin time between 1.5 and 2 times the normal value. The lower speed flow necessary for adequate tissue perfusion is wanted.

Ventilator settings, end-tidal PCO2 monitoring, blood gas analysis and transpulmonary blood flow monitoring

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation and PVA-ECMO support with low residual native cardiac output

Exclusion Criteria:

* age less than 18 years
* pulmonary disorders with abnormal dead-space (obstructive pulmonary disease; acute respiratory distress syndrome)
* cardiac shunt (atrial or ventricular communication)
* significant tricuspid or pulmonary valve disease
* pulmonary artery catheter implantation contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under mechanical ventilation and PVA-ECMO support
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Assessment of end-tidal pressure CO2 (PetCO2) correlation with pulmonary artery flow | Up to 5 days
  end-tidal pressure CO2 (PetCO2) vs pulmonary artery flow measured by pulmonary catheter or echocardiography

SECONDARY OUTCOMES:
Assessment of end-tidal pressure CO2 (PetCO2) thresholds to detect pulmonary artery flow < 1 l/min and indexed flow < 1l/min/m2 | Up to 5 days
Assessment of Factors of end-tidal pressure CO2 (PetCO2) variation | Up to 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- JACOB, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
unkown

REFERENCES:
- [Derived] Mourad M, Eliet J, Zeroual N, Saour M, Sentenac P, Manna F, Molinari N, Gandet T, Colson PH, Gaudard P. Pulse pressure and end-tidal carbon dioxide for monitoring low native cardiac output during veno-arterial ECLS: a prospective observational study. Crit Care. 2020 Sep 22;24(1):569. doi: 10.1186/s13054-020-03280-z. PMID 32962727